CLINICAL TRIAL: NCT04016675
Title: Long-term Outcomes of Neoadjuvant Radiotherapy Versus Adjuvant Radiotherapy for Malignant Lacrimal Sac Tumors (A Multicenter Randomized Controlled Trial)
Brief Title: Neoadjuvant Radiotherapy for Malignant Lacrimal Sac Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Peking University Third Hospital (Other); Tianjin Medical University Eye Hospital (Other); Peking University Eye Center (Other)
Responsible Party: Principal Investigator, Jiang Qian, Professor, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FD-EENT-20190701
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Malignant Tumor of Lacrimal Drainage Structure
MeSH Terms: interventions — Neoadjuvant Therapy; Chemoradiotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Neoadjuvant Radiotherapy/Chemoradiotherapy Followed by Surgery
  Interventions: Other: Neoadjuvant Radiotherapy/Chemoradiotherapy Followed by Surgery
- Control Group (Active Comparator): Surgery Followed by Adjuvant Radiotherapy/Chemoradiotherapy
  Interventions: Other: Surgery Followed by Adjuvant Radiotherapy/Chemoradiotherapy

INTERVENTIONS:
Other: Neoadjuvant Radiotherapy/Chemoradiotherapy Followed by Surgery — After assigned into the study group, subjects will be conducted with incisional biopsy. Based on the tumor type and tumor stage, subjects will be conducted with neoadjuvant radiotherapy/chemoradiotherapy followed by radical surgery and simultaneous orbital reconstruction. After surgery, adjuvant chemotherapy will be determined based on the tumor histology, local tumor invasiveness, proximity of the surgical margins from the tumor, and pronouncement of tumor margins on permanent section tissue review.
  Arms: Study Group
Other: Surgery Followed by Adjuvant Radiotherapy/Chemoradiotherapy — After assignment into the control group, subjects will receive radical surgery without simultaneous orbital reconstruction. Adjuvant radiotherapy / chemoradiotherapy will initiate within two weeks after surgery. Both the radiotherapy and chemoradiotherapy should be comparable between the study group and the control group when tumor characteristics in these two groups are identical.
  Arms: Control Group

SUMMARY:
The treatment for malignant lacrimal sac tumors is difficult and the prognosis is poor. The conventional strategy is surgical resection followed by adjuvant radiotherapy with or without concurrent chemotherapy. This approach has many drawbacks including positive surgical margins due to large tumor size, distant metastasis due to intraoperative squeeze, and implant exposure due to high doses of radiation. In previous research, the investigators innovatively adopted neoadjuvant radiotherapy (or chemoradiotherapy) and withdrew radiotherapy after surgery. Preoperative radiotherapy can effectively reduce the tumor size and encapsulate the tumor in a fibrotic cyst, and therefore enables en-bloc excision of the tumor and simultaneous orbital reconstruction. This multidisciplinary approach can reduce the risk of recurrence and metastasis, lower the dose of radiation, and avoid implant exposure after reconstruction.

In order to compare the long-term outcomes between neoadjuvant radiotherapy and conventional treatment approach, the investigators will prospectively recruit 94 patients with malignant lacrimal sac tumors and randomly assign these subjects into the study group (neoadjuvant radiotherapy, 47 cases) and the control group (conventional treatment, 47 cases). The primary outcomes include overall survival, disease-free survival, distant metastasis-free survival, and locoregional control at 2-year, 5-year and 10-year intervals. The secondary outcomes include ocular functions (visual acuity and diplopia, tear film stability and tear secretion, globe dystopia and motility, and corneal topography), acute and chronic radiation-related toxicity, cosmesis (medial canthal tendon dystopia and eyelid retraction), and assessment of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suggestive symptoms, signs, imaging features and/or biopsy results for malignant lacrimal sac tumors
* Regardless of previous operations including silicone tube intubation, endoscopic dacryocystorhinostomy and incisional/needle biopsy

Exclusion Criteria:

* Recurrent tumors
* Metastatic tumors to the lacrimal sac region
* Malignant lacrimal sac tumors with previous surgical excision
* Malignant lacrimal sac tumors with local nodal or distant metastasis
* Special tumor types (e.g. lymphoma) which require non-surgical treatment
* Large tumors (invades ≥ 2/3 depth of the orbit) which require orbital exenteration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival at 2-year interval | 2 years
  living subjects
overall survival at 5-year interval | 5 years
  living subjects
overall survival at 10-year interval | 10 years
  living subjects
disease-free survival at 2-year interval | 2 years
  tumor-free subjects
disease-free survival at 5-year interval | 5 years
  tumor-free subjects
disease-free survival at 10-year interval | 10 years
  tumor-free subjects
distant metastasis-free survival at 2-year interval | 2 years
  living subjects with no distant metastasis
distant metastasis-free survival at 5-year interval | 5 years
  living subjects with no distant metastasis
distant metastasis-free survival at 10-year interval | 10 years
  living subjects with no distant metastasis
locoregional control at 2-year interval | 2 years
  living subjects without local recurrence or local metastasis
locoregional control at 5-year interval | 5 years
  living subjects without local recurrence or local metastasis
locoregional control at 10-year interval | 10 years
  living subjects without local recurrence or local metastasis

SECONDARY OUTCOMES:
Visual Acuity | up to 2 years
  Best-corrected visual acuity (BCVA) will be measured under standardized lighting conditions in the room, and will be converted to logarithm of the minimum angle of resolution (logMAR) values for statistical analysis.
Subjective Diplopia After Surgery | up to 2 years
  Subjective diplopia will be assessed by categorizing patients according to four grades: no diplopia (absent), diplopia when the patient is tired or awakening (intermittent), diplopia at extremes of gaze (inconstant), and continuous diplopia in the primary or reading position (constant). A change of one grade is considered to be clinically relevant.
Number of Participants with Acute Radiation-Related Toxicity | 1 month
  Acute radiation-related toxicity is defined as events occurring within 1 month after start of radiotherapy, and will be prospectively graded by the treating radiation oncologist according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5).
Number of Participants with Chronic Radiation-Related Toxicity | up to 2 years
  Chronic radiation-related toxicity is defined as events occurring or persisting > 3 months after start of radiotherapy, and will be prospectively graded by the treating radiation oncologist according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5).
Health-Related Quality of life | up to 10 years
  The health-related quality of life will be assessed based on the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Core 30 (QLQ-C30) downloaded from https://www.eortc.org. This 30-item questionnaire includes five functional scales, three symptom scales, a global health status / QoL scale, and six single items. The multi-item scales include a different set of items. Each item includes four subscales, namely "Not at all" (1 point), "A little" (2 points), "Quite a bit" (3 points) and "Very much" (4 points).
  The score will be recorded during each follow-up, and data will be analyzed for comparison between the study group and the control group.
Ophthalmic Cancer-Related Quality of life | up to 10 years
  The ophthalmic cancer-related quality of life will be assessed based on the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Ophthalmic Cancer Module 30 (QLQ-OPT30) downloaded from https://www.eortc.org. The QLQ-OPT30 comprises of 30 questions assessing vision impairment (9 items), functional problems due to vision impairment (8 items), eye symptoms (6 items), worry about recurrent disease (2 items), problems with appearance (1 items), problems driving (2 items), headache (1 item), problems reading (1 item). Each item includes four subscales, namely "Not at all" (1 point), "A little" (2 points), "Quite a bit" (3 points) and "Very much" (4 points).
  The score will be recorded during each follow-up, and data will be compared between the study group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Qian, MD, Study Chair — Fudan Eye & ENT Hospital
Locations (1):
- Fudan Eye & ENT Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes